CLINICAL TRIAL: NCT01278966
Title: Modified Atkins Diet in Children and Adolescents With Drug-resistant Epilepsy - a Prospective Pilot Trial
Brief Title: Modified Atkins Diet in Children and Adolescents With Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Kathrine Haavardsholm, Oslo University Hospital, Division of Surgery and Clinical Neuroscience, National Centre for Child Epilepsy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-09180a (REK)
Record Dates: First submitted 2010-12-29; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; Diet; the Modified Atkins Diet; Ketogenic diet
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Modified Atkins Diet (Experimental): Treatment with the Modified Atkins Diet for 6 months
  Interventions: Other: The Modified Atkins Diet

INTERVENTIONS:
Other: The Modified Atkins Diet — The Modified Atkins Diet; 10 g carbohydrate per day and a high fat intake
  Other Names: Ketogenic diet

SUMMARY:
The purpose of the study is to evaluate the effect of the Modified Atkins Diet in children and adolescents with drug-resistant epilepsy regarding seizure control, and to create a protocol for the use of the Modified Atkins Diet as a treatment for epilepsy in Norway.

DETAILED DESCRIPTION:
The study is a prospective trial on the Modified Atkins Diet for children and adolescents with drug-resistant epilepsy. The Modified Atkins Diet is a less restrictive diet than the classical ketogenic diet, which is usually offered to this group of patients. Twenty patients between 2 and 18 years are included in the study, and the study period is 6 months. The study will be conducted at the National Centre for Child Epilepsy in Norway.

ELIGIBILITY:
Inclusion Criteria:

* age: 2-18 years
* At least 3 epileptic seizures per week
* Tried at least two anti-epileptic drugs without satisfactory seizure control
* Willing to try diet treatment for 6 months

Exclusion Criteria:

* Too difficult for the family to adhere to a strict diet
* Not able to fill in a seizure calendar
* Local authorities will not approve the treatment
* VNS stimulator the last 12 months or changes made to VNS stimulator during the last three months
* Other disease where a diet high in fat is contra indicated
* Diet treatment is not possible because of poor intake of food or fluids
* Cortisol or other medication that influence energy metabolism or epileptic drug metabolism last month
* Patient has the last month used alternative medicine which may influence the diet
* Patient has tried the ketogenic fiet og Modified Atkins diet the last three years
* pregnancy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | 6 months
  Seizure frequency is assessed after 1 month, 3 months and 6 months.

SECONDARY OUTCOMES:
Ambulatory EEG | After 6 months
  24-hours EEG before diet treatment and after 6 months on the diet.
Body Weight | 6 months
  Body weight was measured before diet treatment, after 1 month, 3 months and 6 months.
Quality of life | 6 months
  Questionnaire assessing quality of life and life on a strict diet, assessed after one, three and six months.
Ketosis | 6 months
  Ketosis in blood and urine measured during the whole study period
Dietary records | 10 weeks
  3-days dietary records were obtained after two and ten weeks on the diet.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lossius, Phd, Study Chair — Oslo University Hospital
Locations (1):
- The National Centre for Child Epilepsy, Pb. 53, Bærum Postterminal, Norway